CLINICAL TRIAL: NCT05894239
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Inavolisib in Combination With Phesgo Versus Placebo in Combination With Phesgo As Maintenance Therapy After First Line Induction Therapy in Participants With PIK3CA-Mutated HER2-Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Inavolisib in Combination With Phesgo Versus Placebo in Combination With Phesgo in Participants With PIK3CA-Mutated HER2-Positive Locally Advanced or Metastatic Breast Cancer
Acronym: INAVO122
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO44263; 2022-502046-28-00 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2023-05-24; First posted 2023-06-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Induction Therapy: Phesgo plus Taxane-Based Chemotherapy (Other): Participants will be administered the treatments as outlined in the interventions section.
  Interventions: Drug: Phesgo; Drug: Taxane-based Chemotherapy
- Maintenance Therapy: Inavolisib plus Phesgo (Experimental): Participants will be administered the treatments as outlined in the interventions section.
  Interventions: Drug: Inavolisib; Drug: Phesgo; Drug: Optional Endocrine Therapy of Investigator's Choice
- Maintenance Therapy: Placebo plus Phesgo (Active Comparator): Participants will be administered the treatments as outlined in the interventions section.
  Interventions: Drug: Phesgo; Drug: Placebo; Drug: Optional Endocrine Therapy of Investigator's Choice

INTERVENTIONS:
Drug: Inavolisib — Participants will receive an inavolisib tablet to be taken orally (PO), once a day (QD), on Days 1-21 of each 21-day cycle, beginning on Day (D) 1 of Cycle (C) 1 of maintenance treatment.
  Arms: Maintenance Therapy: Inavolisib plus Phesgo
Drug: Phesgo — Phesgo will be administered to participants subcutaneously every 3 weeks (Q3W) on D1 of each 21-day cycle.
Drug: Placebo — Inavolisib-matching tablet taken PO QD on Days 1-21 of each 21-day cycle, beginning on D1 C1 of maintenance treatment.
  Arms: Maintenance Therapy: Placebo plus Phesgo
Drug: Taxane-based Chemotherapy — During the induction therapy phase, the investigator's choice of taxane-based chemotherapy will be administered after Phesgo.
  Other Names: non-investigational medicinal product (NIMP)
  Arms: Induction Therapy: Phesgo plus Taxane-Based Chemotherapy
Drug: Optional Endocrine Therapy of Investigator's Choice — Optional endocrine therapy (ET) is allowed at the discretion of the investigator, based on the standard of care. Allowed ETs are tamoxifen, or one of the specified third-generation aromatase inhibitor (AI [anastrozole, letrozole, or exemestane]), or fulvestrant. The investigator will determine and supply the appropriate luteinizing hormone-releasing hormone (LHRH) agonist locally approved for use in breast cancer. The LHRH agonist will be administered according to local prescribing information.
  Other Names: NIMP
  Arms: Maintenance Therapy: Inavolisib plus Phesgo; Maintenance Therapy: Placebo plus Phesgo

SUMMARY:
This study will evaluate the efficacy and safety of inavolisib in combination with Phesgo (pertuzumab, trastuzumab, and rHuPH20 injection for subcutaneous use) compared with placebo in combination with Phesgo, as maintenance therapy, after induction therapy in participants with previously untreated HER2-positive advanced breast cancer (ABC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Histologically or cytologically confirmed and documented adenocarcinoma of the breast with metastatic or locally advanced disease not amenable to curative resection
* Confirmation of HER2 biomarker eligibility based on valid results from central testing of tumor tissue documenting HER2-positivity
* Confirmation of PIK3CA-mutation biomarker eligibility based on valid results from central testing of tumor tissue documenting PIK3CA-mutated tumor status
* Disease-free interval from completion of adjuvant or neoadjuvant systemic non-hormonal treatment to recurrence of >= 6 months
* LVEF (left ventricular ejection fraction) of at least 50% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* Adequate hematologic and organ function prior to initiation of study treatment

Exclusion Criteria:

* Prior treatment in the locally advanced or metastatic setting with any PI3K, AKT, or mTOR inhibitor or any agent whose mechanism of action is to inhibit the PI3K-AKT-mTOR pathway
* Any prior systemic non-hormonal anti-cancer therapy for locally advanced or metastatic HER2-positive breast cancer prior to initiation of induction therapy
* History or active inflammatory bowel disease
* Disease progression within 6 months of receiving any HER2-targeted therapy
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Participants with active HBV infection
* Clinically significant and active liver disease, including severe liver impairment, viral or other hepatitis, current alcohol abuse, or cirrhosis
* Symptomatic active lung disease, including pneumonitis or interstitial lung disease
* Any history of leptomeningeal disease or carcinomatous meningitis
* Serious infection requiring IV antibiotics within 7 days prior to Day 1 of Cycle 1
* Any concurrent ocular or intraocular condition that, in the opinion of the investigator, would require medical or surgical intervention during the study period to prevent or treat vision loss that might result from that condition
* Active inflammatory or infectious conditions in either eye or history of idiopathic or autoimmune-associated uveitis in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2032-12-28 (Estimated)

PRIMARY OUTCOMES:
Investigator-Assessed Progression-Free Survival (PFS) | Up to approximately 40 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 111 months
Investigator-Assessed Objective Response Rate (ORR) | Up to approximately 111 months
Investigator-Assessed Duration of Response (DOR) | Up to approximately 111 months
Investigator-Assessed Clinical Benefit Rate (CBR) | Up to approximately 111 months
Investigator-Assessed PFS2 | Up to approximately 111 months
Mean and Mean Changes from Baseline Score in Function and Health-Related Quality of Life (HRQoL) | Day 1 of Cycles 1 and 2 and beyond, 30-day safety follow up visit, post-treatment tumor assessment follow-up with PRO collection and survival follow up visit every 6 months (up to 111 months). Each cycle is 21 days.
  Assessed through the use of the Functional (Role, Physical) and Global Health Status (GHS)/Quality of Life (QoL) scales of the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30)
Percentage of Participants with Adverse Events | Day 1 until 30 days after the final dose of study treatment (up to approximately 111 months). Each cycle is 21 days.
Plasma Concentration of Inavolisib at Specified Timepoints | Day 1 of Cycles 1 and 4. Each cycle is 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (184):
- United States (20):
  - Banner Health MD Anderson AZ, Gilbert, Arizona
  - Disney Family Cancer Center, Burbank, California
  - City of Hope, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Ellison Institute of Technology, Los Angeles, California
  - Georgetown Uni Hospital, Washington D.C., District of Columbia
  - Medstar Research Institute, Hyattsville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atrium Health, Charlotte, North Carolina
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Renovatio Clinical - El Paso, El Paso, Texas
  - JPS Health Network, Fort Worth, Texas
  - Lumi Research, Kingwood, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Swedish Medical Center, Seattle, Washington
- Argentina (6):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
  - Instituto de Oncología de Rosario, Rosario
  - Hospital Provincial del Centenario, Rosario
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Clínica Viedma, Viedma Rio Negro
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Monash Health, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - CHIREC, Auderghem
  - CHU Brugmann (Victor Horta), Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Les Viviers, Charleroi
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - Clinique Ste-Elisabeth, Namur
- Brazil (11):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor Amazônia, Porto Velho, Rondônia
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Canada (9):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - The Moncton Hospital, Moncton, New Brunswick
  - Eastern Health - General Hospital, St. John's, Newfoundland and Labrador
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier de l?Université de Montréal (CHUM), Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
  - Allan Blair Cancer Center, Regina, Saskatchewan
- China (16):
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sichuan Provincial Cancer Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Tumor Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - The First Affiliated Hospital to Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Shantou Center Hospital, Shantou
  - Tianjin Cancer Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
- Colombia (4):
  - Clinica De La Costa, Barranquilla
  - Fundación CTIC - Centro de Tratamiento e Investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogota, D.C.
  - Oncomedica S.A., Montería
  - Sociedad de Oncología y hematología del Cesar Ltda, Valledupar
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku Uni Central Hospital, Turku
- France (5):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
- Germany (12):
  - Klinikum St. Marien, Amberg
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Marienhospital Bottrop gGmbH, Bottrop
  - Gynonco Düsseldorf, MVZ Medical Center GmbH, Düsseldorf
  - Frauenarztpraxis Dr. Apel, Dr. Kolpin, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Klinik & Poliklinik für Frauenheilkunde und Geburtshilfe, Campus Innenstadt, München
  - St. Franziskus Hospital Münster;Studiensekretariat der onkologischen Zentren, Münster
  - Caritas Klinik St. Theresia -Frauenklinik Brustzentrum, Saarbrücken
  - Gynäkologie Kompetenzzentrum, Stralsund
  - Universitätsfrauenklinik Ulm, Ulm
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- India (7):
  - Gujarat Cancer & Research Inst., Ahmedabad, Gujarat
  - Sunshine Global Hospital (A unit of Baroda Medicare Pvt Ltd), Surat, Gujarat
  - Artemis Hospital, Gurugram, Haryana
  - Sir H. N. Reliance Foundation Hospital and Research Centre, Mumbai, Maharashtra
  - National Cancer Institute, Nagpur, Maharashtra
  - Max Super Speciality Hospital, NEW Delhi Delhi, National Capital Territory of Delhi
  - Tata Medical Center, Kolkata, West Bengal
- Italy (10):
  - I.R.S.T Srl IRCCS, Meldola, Emilia-Romagna
  - Ospedale San Giovanni Addolorata, Rome, Lazio
  - Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Casa di Cura La Maddalena, Palermo, Sicily
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, Tuscany
  - "Azienda Ospedaliera Universitaria Integrata Verona Ospedale Borgo Trento", Verona, Veneto
- Japan (2):
  - Chiba Cancer Center, Chiba
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
- King Hussein Cancer Center, Amman, Jordan
- University of Nairobi - Institute of Tropical and Infectious Diseases, Nairobi, Kenya
- Mexico (5):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - OncoMed, Mexico City, Mexico CITY (federal District)
  - Centro Oncológico Hematológico Roma, Mexico City, Mexico CITY (federal District)
  - Hospital Universitario, Monterrey, Nuevo León
  - CENEIT Oncologicos, Mexico City
- Sultan Qaboos Comprehensive Cancer Care & Research Center, Muscat, Oman
- Poland (8):
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Szpital Morski im.PCK, Gdynia
  - Narodowy Instytut Onkologii Odzia? w Gliwicach, Gliwice
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Wielkopolskie Centrum Onkologii im. Marii Sk?odowskiej-Curie, Późna
  - Centrum Onkologii Instytut im.M. Sklodowskiej-Curie, Warsaw
- Singapore (4):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Icon Cancer Centre Farrer Park, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (6):
  - Hopelands Cancer Centre, Hilton
  - Charlotte Maxeke Academic Hospital, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Limpopo Cancer Research Institute, Polokwane
  - Steve Biko Academic Hospital, Pretoria
  - Chris Hani Baragwanath Clinical Trial Site, Soweto
- South Korea (7):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (3):
  - National Taiwan Uni Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou, Taoyuan
- Tunisia (5):
  - Abderrahmen Mami Hospital, Aryanah
  - Taher Maamouri Hospital, Nabeul
  - Habib Bourguiba Hospital, Sfax
  - Farhat Hached Hospital, Sousse
  - Institut Salah Azeiz, Tunis
- Turkey (Türkiye) (9):
  - Sakarya Training and Research Hospital, Adapazarı
  - Gulhane Training and Research Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Dicle University Faculty of Medicine, Diyarbakır
  - Medipol Mega Üniversite Hastanesi Göztepe, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Medical Park Seyhan Hospital, Seyhan
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara
- Uganda Cancer Institute, Kampala, Uganda
- United Kingdom (6):
  - Belfast City Hospital, Belfast
  - Blackpool Victoria Hospital, Blackpool
  - Colchester General Hospital, Colchester, Essex
  - Mount Vernon Hospital, Northwood
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing